CLINICAL TRIAL: NCT04516252
Title: A Health-literacy Module for Overweight Adolescents and Their Parents on Canine Physical Activity, Nutrition and Behavior: Enhancing Department of Health and Human Services' (DHHS) BodyWorks Program At a Federally Qualified Health Center
Brief Title: Enhancing BodyWorks: a Canine Health Literacy Module
Acronym: BW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of Southern California (Other); Tufts Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Larry Yin, Associate Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHLA-CG-19-00001; R21HD097761 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-18 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Overweight and Obesity; Overweight Adolescents
Keywords: Overweight; Obesity; children; adolescents; comprehensive family lifestyle intervention program; telehealth; BodyWorks; Human Animal Interaction
MeSH Terms: conditions — Overweight; Obesity; Human-Animal Interaction | interventions — Ecological Momentary Assessment; Fitness Trackers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Half of the BodyWorks families will be randomized to the intervention group, and will receive a PAT for the children, the parents, and the dogs at the beginning of the cycle; the children will respond to EMA surveys using a cell phone; the children and the parents will receive the Canine health literacy module in addition to the BW curriculum.
  Interventions: Behavioral: BodyWorks Intervention; Behavioral: Canine Curriculum; Behavioral: Ecological Momentary Assessment; Behavioral: Physical Activity Trackers
- Control (Active Comparator): Half of the BodyWorks participants will be randomized to the control group and will receive a PAT at the beginning of the cycle for the children, the parents, and the dogs, and the children will respond to EMA surveys using cell phones.
  Interventions: Behavioral: BodyWorks Intervention; Behavioral: Ecological Momentary Assessment; Behavioral: Physical Activity Trackers

INTERVENTIONS:
Behavioral: BodyWorks Intervention — BodyWorks (BW), a Comprehensive Behavioral Family Lifestyle Interventions (CBFLI), a national, empirically validated, curriculum-based 7-week program will be implemented (Borden et al., 2012; DHHS, 2013)
Behavioral: Canine Curriculum — Using our team's expertise in veterinary medicine, human-animal interaction, and animal behavior modification, develop an empirically-based, 7-week module on canine health and behavior.
  Arms: Intervention
Behavioral: Ecological Momentary Assessment — Ecological Momentary Assessments (EMA) of physical activity will be conducted using mobile phones for 7 weeks of the BW program, prospectively collecting data on 4 days per week (Saturday to Tuesday) (Dunton et al., 2011; Liao et al., 2016).
Behavioral: Physical Activity Trackers — Three types of consumer-grade wireless personal activity trackers (PATs): FitBit Inspire® designed for children 8 years of age and older; FitBit Inspire® for adults (Diaz et al., 2015; Espinoza et al., 2017); and FitBark®, wireless, global positioning systems (GPS)-based personal activity trackers for dogs (Patel et al., 2017). This approach will allow us to evaluate quantity (number of steps) and intensity of physical activity in the adolescents, their parents, and their dogs, as well as to synchronize Fitbit Ace and FitBark to establish the amount of shared physical activity of adolescents and their dogs.

SUMMARY:
Dog ownership can serve as a vehicle for large-scale multi-level public health interventions, especially for pediatric overweight and obesity, due to dogs' unique place in children and adolescents' social networks.This study develops and tests a novel approach to design a Canine Health-Literacy module to enhance a Comprehensive Family Lifestyle Intervention BodyWorks, for dog-owning adolescents who have been diagnosed with overweight or obesity, and their parents. The results are anticipated to make an important step towards addressing the overweight and obesity epidemic among both people and companion dogs in the U.S.

DETAILED DESCRIPTION:
This project is a feasibility, acceptability, and pilot study that leverages the psychosocial benefits of informed and attached dog ownership among treatment-naïve overweight or obese adolescents. It is based upon a socioecological model of health behavior that pursues multiple levels of influence, including those extending across species lines such as physical activity. BodyWorks, a Comprehensive Behavioral Family Lifestyle Interventions (CBFLI), a national, empirically validated, curriculum-based 8-week program (orientation and 7 weeks of curriculum) will be offered at Children's Hospital Los Angeles AltaMed Division of General Pediatrics, a Federally Qualified Healthcare Center. The aims of the study are: Specific Aim 1: Using current empirical evidence in veterinary medicine, to develop a Canine Health Literacy module (CHL) to be delivered as part of the existing, empirically tested BW curriculum to increase adolescents' health literacy about their dogs' physical activity needs, weight status, and nutrition. Specific Aim 2: Test the feasibility and acceptability of a concurrent approach using physical activity trackers and Ecological Momentary Assessment. 2(a): Test the feasibility and acceptability of objective measurement of physical activity using wireless fitness trackers for adolescents (FitBit Inspire), their parents (FitBit Inspire), and their dogs (FitBark); 2(b): Test the feasibility and acceptability of using mobile phones for Ecological Momentary Assessment of types and contexts of adolescent's physical activity with dogs. Specific Aim 3: To establish the size of the effect, and the variability associated with the 8 week-long BW + CHL module, as compared with the control group who received the standard BW program in 3(a) adolescents' positive affect during or after physical activity with the dog, as measured by the Ecological Momentary Assessment using prompts on mobile phones; and 3(b) levels of overall physical activity for the adolescents, their parents, and the dogs as measured by the FitBit Ace (adolescents), FitBit Flex2 (parents), and FitBark (dogs). The project will establish feasibility, acceptability, attrition, and protocol compliance, and will collect pilot data needed for power calculations in preparation for an R01 Randomized Controlled Trial as a next step to test the effectiveness of our enhanced BW+CHL program. This project represents a significant methodological and theoretical advancement in the field of Human-Animal Interaction (HAI) and in research on overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese youth ages 9-17 years and their caregivers
* Own dog

Exclusion Criteria:

* Normal BMI
* Do not own dog

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Estimated)
Dates: Start 2021-02-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Variability associated with the BodyWorks + Canine Health Literacy intervention | Change from baseline physical activity at 7 weeks
  Determining the mean difference between groups in the physical activity outcomes for number of steps per day as measured by the physical activity tracker
Affect Variability associated with the BodyWorks + Canine Health Literacy intervention | Change from baseline affect at 7 weeks
  Determining the mean difference between the groups in the positive and negative affect ecological momentary assessment outcomes.
Feasibility of Ecological Momentary Assessment | Weeks 1, 4, 7 of intervention
  Feasibility will be determined by data completeness: Ratio of questions answered during a wave to total number of possible questions.
Acceptability of Ecological Momentary Assessment | Week 7 of intervention
  Acceptability will be measured by EMA prompt response rate out of the total possible responses.
Feasibility of use of physical activity trackers | Weeks 1-7 of intervention
  Feasibility will be determined by data completeness: Ratio of days on which there are valid fitbit data out of the total number of days in terms of steps per day and minutes per day.
Acceptability of use of physical activity trackers | Week 7 of intervention
  Acceptability will be measured by response rate on user satisfaction survey.
Physical activity for adolescents | daily for 7 weeks
  Number of steps per day
Physical activity for parents | daily for 7 weeks
  Number of steps per day
Physical activity for dogs | daily for 7 weeks
  Number of steps per day
Ecological Momentary assessments of adolescents | Weeks 1, 4, 7
  Mean adolescent affect ratings measured by ecological momentary assessments administered via text messages

SECONDARY OUTCOMES:
Body Mass index | Change from baseline BMI at 7 weeks
  Weight and height will be used to calculate BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Larry Yin, MD, MSPH, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- AltaMed@CHLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No